CLINICAL TRIAL: NCT05854927
Title: Impact of the Spatial Resolution of Several Contrast-enhanced 3D T1-WI Sequences When Diagnosing Giant Cell Arteritis (GCA)
Acronym: SPARTA
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2022_14
Record Dates: First submitted 2023-04-27; First posted 2023-05-11 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 3D T1 MRI sequences injected with fat saturation and black blood — 3D T1 MRI sequences injected with fat saturation and black blood

SUMMARY:
Giant cell arteritis (GCA) (or Horton's disease) is a segmental and focal inflammatory arteritis affecting large and medium-sized arteries. Its incidence is estimated at 17.8/100,000 in subjects over 50 years old (and 46/100,000 in subjects over 70 years old). This disease remains a severe pathology due in particular to its vascular, ophthalmological, neurological, cardiac and aortic complications. In case of suspected CAG, management is a real therapeutic emergency. Indeed, only corticosteroid therapy started as early as possible can prevent the occurrence of these complications.

The gold standard for the diagnosis of CAG has long been the temporal artery biopsy, but imaging is now considered as a 1st line diagnostic examination for the diagnosis of CAG according to the EULAR 2018 recommendations. Notably, temporal artery MRI has excellent sensitivity and specificity for diagnosis.

However, the high diagnostic performance of MRI has been achieved by performing 3D T1 black blood and fat saturation sequences in high resolution (<0.7mm), which are not accessible in all centers in France and worldwide.

The realization of identical sequences with a lower resolution could allow a greater generalization of these sequences and improve the diagnostic management of GCA patients, including in non-expert centers.

The objective of our study is to investigate the diagnostic performance of several 3D T1 black blood and fat saturation sequences for the diagnosis of GCA.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Referred for imaging for an injected MRI for suspected GCA
* Suspicion of GCA based on the presence of three major criteria or two major and one minor criteria defined as follows:

  * Major criteria: Age > 50 years; Headache of recent onset; Claudication of the jaw, tongue or swallowing disorders; Visual problems (blindness, diplopia, blurred vision - including visual accidents occurring during the first week of treatment); Sedimentation rate at 1st hour > 50 and/or CRP > 8mg/l
  * Minor criteria: Hypersensitivity or induration of the scalp or presence of nodules remote from the temporal artery; Temporal artery abnormalities on palpation; Facial pain or feeling of facial edema; General signs (fever >38°C, weight loss >10%, anorexia, malaise, asthenia).
* Cconsent to participate in the study
* Affiliated or beneficiary of a social security plan

Exclusion Criteria:

* Newly diagnosed malignant disease (diagnosed less than one year prior to inclusion)
* Active infectious disease
* Autoimmune disease (especially but not limited to: Wegener's disease, Takayasu vasculitis, ANCA vasculitis, rheumatoid arthritis, lupus erythematosus, periarteritis nodosa).
* Systemic corticosteroid therapy for more than 10 days at high dose (>0.5mg/kg/d of prednisone)
* Contraindication to MRI
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation in the study will be offered to all patients referred to imaging for an injected MRI for suspected GCA.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of unilateral or bilateral inflammation of the temporal arteries and/or ophthalmic arteries or other branch of the internal carotid arteries with a 3D PDw MRI sequence for GCA diagnosis | Month 3
  The gold standard for the diagnosis of GCA will be based on a multidisciplinary evaluation (internists, neurologists, ophthalmologists) of the clinical and biological data in the patient's file at 3 months of inclusion, according to the criteria of the ACR (American College of Rheumatology) 2021, blinded to the MRI scans performed at inclusion.
  MRI imaging will be reviewed by two radiologists (one junior and one senior) to assess inflammation in each artery of interest. Consensus will be sought in the event of disagreement between the two readers.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France